CLINICAL TRIAL: NCT03214770
Title: Antibacterial Effect of Light-activated Calcium Silicate Versus Calcium Hydroxide on Permanent Carious Molars Treated With Step-wise Excavation (A Randomized Clinical Trial)
Brief Title: Antibacterial Effect of Light-activated Calcium Silicate Versus Light-activated Calcium Hydroxide
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Morsy Mohamed, Master student at conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: oper 246
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Dental Caries Extending Into Dentin
MeSH Terms: interventions — TheraCal; Biner LC

STUDY DESIGN:
Who Masked: Participant
Masking Description: It will be a single-blinded study so that the participant will be blinded, the researcher and the data analysis will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Light-cured calcium silicate (Experimental): This biomaterial calcium silicate is manufactured to have an anti-bacterial effect on micro-organisms within the dentin, thus allowing the inhibition of bacterial growth therefore no caries will progress. Material is injected and light-cured within the dentin and sealed with a restoration.
  Interventions: Drug: TheraCal
- Light-cured calcium hydroxide (Active Comparator): This biomaterial calcium hydroxide is manufactured to have an anti-bacterial effect on micro-organisms within the dentin, thus allowing the inhibition of bacterial growth therefore no caries will progress. Material is injected and light-cured within the dentin and sealed with a restoration.
  Interventions: Drug: light-cured calcium hydroxide

INTERVENTIONS:
Drug: TheraCal — Biomaterial used for carious lesions reaching to dentin. Material is applied and after 6 month dentin sample collection and the bacterial count by digital colony counter, Agar diffusion test.
  Other Names: light-cured calcium silicate
  Arms: Light-cured calcium silicate
Drug: light-cured calcium hydroxide — Biomaterial used for carious lesions reaching to dentin. Material is applied and after 6 month dentin sample collection and the bacterial count by digital colony counter, Agar diffusion test.
  Other Names: Biner LC
  Arms: Light-cured calcium hydroxide

SUMMARY:
This is a randomized clinical study. 48 subjects with a confirmed diagnosis of deep carious molars without pulpal lesions were randomized to one of two treatments: Patients treated with Light-cured calcium silicate (Theracal) liner, or treated with light-cured calcium Hydroxide (Biner LC) liner. Both two Treatments are with the step-wise excavation Technique.

Treatment will be done at baseline, collecting dentin sample before application of liner material, then patients will be dismissed with Resin-modified Glass Ionomer restoration and recalled after 6 months. Re-entry of tooth required for completing the step-wise excavation technique collecting the second dentin sample after this time interval (6 months) and permanently restore tooth with composite restoration. Dentin samples will be microbiologically analyzed and the results will be statistically calculated.

DETAILED DESCRIPTION:
1. Study setting:

   This study will be carried out on adult patients attending to the operative clinic in The Faculty of Oral and Dental Medicine, Cairo University, Egypt. The procedures will be carried out by postgraduate student Hanaa Mohamed Morsy [B.D.S. 2011 from Misr University for Science and Technology] without an assistant.
2. Variables of the study: A total of 48 carious lesions will be included in the study. Divided into two groups 24 each. Thus 48 dentin samples will be collected from each group (24 pre-operative dentin sample and 24 dentin sample after 6 months post-operative)
3. Trial Description:

   • Grouping of participants: Patients will be diagnosed to find carious molars reaching dentin level. Participants will be divided to two groups randomly according to the type of liner that will be placed and sample of dentin that will be taken before placement of liner and after placement (6 months); D1 Dentin sample before and after treatment with light-cured Calcium Silicate (Theracal) {n=48}, and D2 Dentin sample before and after treatment with light-cured Calcium Hydroxide ( Biner LC){n=48}.

   • Intervention/ Control: The procedure will be formed by removing the caries tissue till reaching dentin, leaving the deep layer for the application of the step-wise technique. Dentin sample will be taken by a spoon excavator for both groups and stored in a media to be transferred to the microbiological lab for analysis at the time baseline of the study (T1). Liner will be applied in the cavity for Group D1 using Theracal, and D2 using Biner LC. For both two groups, molars will be restored with Glass Ionomer restoration at the time baseline. Patients will be recalled after 6 months for the re-entry of the restored teeth , removing the Glass Ionomer restoration and collect the dentin sample (T2) for evaluation of the microbiological count. Finally restoring the teeth with Composite as the final permanent restoration. the procedure will follow the manufacturer's instructions for every material used.

   • Outcome: The outcome will be the bacterial count of Streptococcus Mutans of the dentin samples collected from the tooth included in the study. Agar Diffusion test and Digital Colony Counter will be conducted for the study. The measuring unit of the bacterial count is CFU/ml. The first dentin sample will be collected in the baseline time and the second dentin sample after 6 month for each group.

   • Randomization: Randomization will be done according to a check list done by a dentist other than the researcher including the number of participants divided into 2 subgroups denoting with letter A, B.

   • Microbiological analysis: Samples will be vortexed for 15 s, diluted, and measured aliquots of the dilutions will be cultivated in duplicate in 3 different culture media. Mitis Salivarius agar supplemented with sucrose and bacitracin will be used for counting of mutans streptococci . For isolation of lactobacilli, Rogosa selective Lactobacillus agar will be used. Counts of total colony forming units (CFU) will be obtained by culture in brain heart infusion agar supplemented with 5% sheep blood and enriched with k-hemin vitamin. The Mitis Salivarius will be incubated under CO 2 conditions at 37 0C for 48 h. Colonies of mutans streptococci will be counted based on their morphology and confirmed with catalase test. Rogosa SL Agar and the BHI will be incubated anaerobically at 37 8C for 72 h. The BHI will be also incubated aerobically at 37 8C for 48 h to determine the total aerobic counts (AE).

   • Sample size calculation: The aim of this study is to evaluate the antibacterial action of TheraCal (light-cured Calcium Silicate base/liner), comparing this material with Calcium Hydroxide paste. If the expected clinical differences in bacterial count by digital colony counter, agar diffusion test is 1± 1. Using power 80% and 5% significance level , we will need to study 17 in each group to be able to reject the null hypothesis that the population means of the experimental and control groups are equal. This number is to be increase to 24 in each group to compensate for possible losses during follow up according to Petrou et al., 2014. The sample size was calculated by PS program.

   • Recruitment: Announcement to residents of outpatient clinic in Conservative Dentistry- Faculty of Oral and Dental Medicine- Cairo University Egypt, to screen adult patient during diagnosis for their chief complain so patients with at least one carious teeth with no pulpal symptoms will be enrolled in this study, if they meet the eligibility criteria.

   • Allocation:
   1. Sequence generation :

      -Randomization is done by computer software www.random.org.

      -The sequence generates 2 codes (A and B). Sample size 24 in each group to compensate for possible losses during follow up.
   2. Allocation and concealment arrangement:

      - A checklist will be designed by a dentist other than the researcher to identify each material specimen
   3. Implementation :

      -Allocation sequence will be generated at the Center of Evidence Based Dentistry, Faculty of Oral and Dental Medicine - Cairo University.

      -Participant enrollment will be done by the principle investigator.

      • Blinding: It will be a single-blinded study so that the participant will be blinded, the researcher and the data analysis will be unblinded.

      • Data collection methods: There will be a file for each participant includes his/her( informed consent, the 2 time interval appointments, all data including address, phone numbers) and all information that will be needed for follow up.
      * Retention:

        -In order to ensure that the participants will come back for the sequence visits, the patient will be asked for the telephone number and address and will be called before the visit.

        -Explanation of the importance of the study is explained to patient and the importance on keeping the appointments.
      * Data management :

        -Explain to the patient the importance of this study and that commitment to the appointments is mandatory to get the best results from this study.
        * All data is documented in the patient sheet.
      * Statistical Methods:

      Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Data will be explored for normality using Kolmogrov-Smirnov test and Shapiro-Wilk test. Comparisons between two groups for normally distributed numeric variables will be done using the Student's t-test while for non normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.( Petrou et al., 2013)

      • Data Monitoring: This study will be monitored by the supervisors who will have full access to the results and will take the final decision to terminate the trial.

      • Harms: No reported adverse effect of the intervention was reported. In case of any harm during the trial it will be reported, documented and treated.

      • Auditing: Auditing of the study design will be done by the evidence based committee- Faculty of Oral and Dental Medicine- Cairo University.
      * Ethics and dissemination:

        -Patient consent.

        -Detailed check list including the exact procedure and intervention that will be performed, the number of visits, the importance of this study to the participants, as well as its importance to the population, and the possible adverse effects accompanied with the use of the intervention.
      * Research ethics approval:

        -This protocol and the template of informed consent form will be reviewed by the Ethics Committee of scientific research, Faculty of Oral and Dental Medicine- Cairo University.
      * Protocol amendments:

        -Any modifications to the protocol which may have an impact on the conduction of the study, potential benefit of the patient or may affect the patient safety, including changes of study objectives, study design, sample size, study procedure or significant administrative aspects will require a formal amendment to the protocol. Such amendment will be agreed upon by the council of Conservative dentistry Department.
      * Consent and assent:

        * Researcher will discuss the trial with the participant's. They will be able to discuss his thoughts with the researcher after a full explanation of the procedure in simple words. A verbal assent will be taken from the participating patient while a written consent is signed by the patient.
      * Confidentiality:

        * All study related information will be stored securely. All participants'' information will be stored in a locked file cabinets in areas with limited access. Process and administrative forms will be identified by a coded ID [identifier number] only to maintain participants' confidentiality. All records that contain names or other personal identifiers will be stored separately from study records identified by code number.
      * Declaration of interest:

      Non-financial

      • Access to data: All principle investigators will be given access to the data sets. All data sets will be password protected.

      • Ancillary and post-trial care: Full mouth treatment will be offered to all the participants in addition to post-operative care and preventive measures after the end of the trial.
      * Dissemination policy:

        1. Trial results:

           -The study results and conclusions are planned to be discussed in the Department of Conservative Dentistry, Faculty of Oral and Dental Medicine, Cairo University through a power point presentation.

           -This study is planned to be published
        2. Authorship:

           -All the authors meet the criteria for authorship which are defined by the International Committee of Medical Journals Editors.
           * Before submission, Trial version will be reviewed and approved by the authors, Evidence-Based Dentistry Committee and Research Ethics Committee at Faculty of Oral and Dental Medicine- Cairo University and screened for plagiarism detector to ensure original work.
           * Role of authors will be declared in details before submission.
           * No professional writers will be used C) Reproducible research The trial reports and full study report will be available.

ELIGIBILITY:
Inclusion Criteria:

1. Normal adults will be recruited in this study, all the volunteers participated in this experiment will be healthy looking with free medical history.
2. Subjects aged between 18-40 years.
3. In each patient required one or two deep carious tooth occlusally either upper or lower permanent molars.
4. All volunteers must be with good oral hygiene in order to restore with composite restorations.
5. Subjects were required to be available for the duration of the study, and to sign an informed consent form

Exclusion Criteria:

1. Subjects with a history of allergy to any of the drugs or chemicals used in the study.
2. Subjects with carious anterior tooth are not within the study.
3. History of pulp pathology of the teeth which indicates root canal treatment is not included in the study.
4. Pregnancy and Lactating mothers.
5. Patients with any systematic problems or mental or physical disability.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-08-10 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial Count | an average of 6 months
  will be done by Digital colony counter, Agar Diffusion Test The measuring unit of the bacterial count is CFU/ml(colony-forming units per milliliter) for liquids). The first dentin sample will be collected in the baseline time and the second dentin sample after 6 month for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Omaima M Safwat, PHD, Study Director — Professor of Conservative Dentistry, Cairo University; Mohsen A Elhassan, PHD, Study Chair — Professor of Conservative Dentistry, Cairo University
Locations (1):
- Hanaa Mohamed Morsy Mohamed, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Petrou MA, Alhamoui FA, Welk A, Altarabulsi MB, Alkilzy M, H Splieth C. A randomized clinical trial on the use of medical Portland cement, MTA and calcium hydroxide in indirect pulp treatment. Clin Oral Investig. 2014;18(5):1383-9. doi: 10.1007/s00784-013-1107-z. Epub 2013 Sep 17. PMID 24043482